CLINICAL TRIAL: NCT04124224
Title: Unidos: Linking Individuals to Social Determinant and Community Health Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: El Rio Community Health Center (Other); Pima County Health Department (Unknown); Yuma County Health District (Unknown); Sunset Community Health Center (Unknown); Maricopa County Health Department (Unknown); Valle del Sol Community Health (Unknown); Mariposa Community Health Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: U48DP006413 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-11 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Chronic Disease; Community Health Workers
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unidos Participants: In the Unidos intervention the county/community-based CHWs will: 1) support and connect participants to health promotion resources; 2) provide individual and group-based support guided by a novel framework for understanding Latino's health advantages, the sociocultural resiliency model; and, 3) leverage community resources to help individuals address SDH-related needs.
  Interventions: Other: Unidos
- Non-Unidos Participants: Comparison Group: Using propensity score matching, the investigators will use the medical records of Unidos participants and the electronic health record comparison group to compare health outcomes.

INTERVENTIONS:
Other: Unidos — The investigators will collaborate with our community partners to implement and evaluate a Community-Clinical Linkage (CCL) model in which Community Health Workers (CHWs) connect individuals to social determinant and community health services and build sociocultural resilience through CHW-facilitated individual and group support. As a public health practice-based study that incorporates evidence-based strategies, the investigators seek to establish Unidos effectiveness in Arizona counties with the highest percentage of Latinos of Mexican origin (Yuma, Pima, Santa Cruz, and Maricopa). Unidos CHWs, based in local health departments, will use evidence-based strategies to address three elements that are important in addressing chronic disease risk: 1) health promotion resources and programs; 2) individual and group-based social support; and 3) leveraging community resources to address social determinants of health.
  Groups: Unidos Participants

SUMMARY:
For 19 years, the Centers for Disease Control and Prevention-funded Arizona Prevention Research Center (AzPRC) has been engaged in academic community collaborative research to reduce chronic disease health disparities among the Latino border communities in Arizona. Our research project, Unidos: Linking Individuals' to Social Determinant and Community Health Services, will result in a model Community-Clinical Linkage intervention to reduce chronic disease risk among Latinos in Arizona. Further, the investigators expect this intervention model to be applicable in other regions and populations. To execute this research, the AzPRC will implement the intervention in partnership with county health departments and Federally Qualified Health Centers. In Unidos the county/community-based CHWs will: 1) support and connect participants to health promotion resources; 2) provide individual and group-based support guided by a novel framework for understanding Latino's health advantages, the sociocultural resiliency model; and, 3) leverage community resources to help individuals address SDH-related needs.

DETAILED DESCRIPTION:
Latinos in Arizona, who are predominantly of Mexican-origin, are disproportionately affected by chronic disease and social conditions that contribute to health disparities. Important social determinants of health (SDH)--conditions where people live, work, and play--include barriers to healthy food, physical activity, poverty, discrimination, and housing instability as well as insufficient access to quality and culturally-responsive services. Such factors are increasingly recognized within primary care and population health as equal drivers of chronic disease and clinical indicators. Latino health is complex with not only disproportionate barriers, but also health advantages compared to other groups.

Recently, federally qualified health centers (FQHCs) have begun to incorporate assessments of their clients' SDH. With their foci on high-level clinical care for underserved populations, however, the capacity of these entities to respond to social and community needs is markedly limited. Community-clinical linkage (CCL) models provide opportunities for FQHCs to work collaboratively with other entities to leverage extant community resources and capacities. County health departments are uniquely positioned to collaborate with primary care partners and other community agencies to address social determinants.

Existing evidence of the effectiveness of CCLs in improving the health status of Latinos and their antecedent social conditions is scarce. The AzPRC will address this gap by executing a practice-based public health research study within four underserved, predominantly Mexican-origin communities. Our core research project, Unidos: Linking Individuals' to Social Determinant and Community Health Services, will result in a model CCL intervention to reduce chronic disease risk among Latinos in Arizona. Further, the investigators expect this intervention model to be applicable in other regions and populations. To execute this research, the AzPRC will implement the intervention in partnership with county health departments and FQHCs. In Unidos the county/community-based CHWs will: 1) support and connect participants to health promotion resources; 2) provide individual and group-based support guided by a novel framework for understanding Latino's health advantages, the sociocultural resiliency model; and, 3) leverage community resources to help individuals address SDH-related needs. The aims of this research study are to

1. Implement and evaluate Unidos, a community-delivered, SDH-focused CHW intervention. The core elements of the evaluation will include community-responsive, mixed methodologies. Our hypothesis is that the Unidos intervention will reduce overall chronic disease risk, defined from the biological component from the American Heart Association's Life's Simple 7. A rigorous quasi-experimental design will be employed to determine Unidos' effect from electronic health records extracted 12 months after enrollment, with comparisons of clients participating vs not participating in the 6-month intervention. Exploratory analyses of cost effectiveness will be executed to further inform the scaling and sustainability of the intervention within local and county health department infrastructures.
2. To test the sociocultural resilience model of Latino health advantages through the collection and analysis of longitudinal data that includes rich markers of reported health status, health behaviors, and psychosocial factors. The investigators have two hypotheses: a) the CHW-led, culturally embedded, intervention will lead to enhanced social support, social networks, health behaviors, quality of life and general health; and b) social support and social networks will mediate improvements in reported health observed over 6 months.
3. A secondary aim is to examine whether our novel, CHW-administered assessments, contribute to the understanding of Latino health risk and advantages beyond a self-administered SDH tool that recently became integrated in the electronic health record (EHR) of two of our four clinical partners. The partners' use of this self-administered SDH tool is part of a national effort where select FQHCs across the country are testing whether it has utility for understanding and better addressing the population health needs of the patients they serve.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 years or older;
* Adults of Latino origin;
* Participants who speak either English or Spanish; and
* Participants who consent to participate in the study.

Exclusion Criteria:

* Excluded will be participants who do not consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Arizona counties with significant Latino populations experience underlying social and economic disparities that place them at risk for chronic disease and negative health outcomes. The participating Maricopa, Pima, Yuma, and Santa Cruz counties are where a significant number of the Latino population for the state reside. Compared to the US population, communities in Arizona with a higher percentages of Latinos are more likely to face poverty, be uninsured, and have chronic disease risks.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Disease Risk | 9 months
  Number of Participants with Chronic Disease Risk as Assessed by the American Heart Association Simple 7 (smoking, nutrition, physical activity, weight, blood pressure, cholesterol, and blood sugar) Change from Baseline in Simple 7 score at 3, 6, and 9 months.
Social Networks | 6 months
  Number of Participants with Improved Social Networks as Assessed by the Berkman-Syme Network Index, Change from Baseline to 6 month follow-up.
Unidos Implementation within Local Health Departments | 2 months
  Organizational readiness as assessed through qualitative data collection including focus groups and interviews.
Social Determinant of Health Factors | 6 months
  Number of participants with improved Social Determinant of Health Factors as assessed by the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences (PRAPARE), change from baseline to 6 month follow-up.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mariposa Community Health Center, Nogales, Arizona
  - Maricopa County Health Department, Phoenix, Arizona
  - Valle del Sol Community Health, Phoenix, Arizona
  - El Rio Community Health Center, Tucson, Arizona
  - Pima County Health Department, Tucson, Arizona
  - Sunset Community Health Center, Yuma, Arizona
  - Yuma County Health District, Yuma, Arizona

IPD SHARING:
Plan to Share IPD: No
As this is a community-based participatory research study, the investigators will work with our Community Action Board to determine what data will be shared.